CLINICAL TRIAL: NCT00928681
Title: A Randomized, Double-Blind (Sponsor Open), Placebo Controlled, Dose Escalating, Parallel Group, Multi-Centre Study To Investigate The Safety, Toleration, Pharmacokinetics And Pharmacodynamics Of Single And Multiple Intravenous/Sub-Cutaneous Doses Of PF-00547659 In Patients With Active Ulcerative Colitis.
Brief Title: A Study To Investigate The Safety And Efficacy Properties Of PF-00547659 In Patients With Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7281001
Record Dates: First submitted 2009-06-22; First posted 2009-06-26 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- 0.03 mg/kg or placebo iv (Other)
  Interventions: Biological: Single dose-group A
- 0.1 mg/kg or placebo iv (Other)
  Interventions: Biological: Single dose-group A; Biological: Multiple dose- Group B
- 0.3 mg/kg or placebo iv (Other)
  Interventions: Biological: Single dose-group A; Biological: Multiple dose- Group B
- 1.0 mg/kg or placebo iv (Experimental)
  Interventions: Biological: Single dose-group A
- 3.0 mg/kg or placebo sc (Other)
  Interventions: Biological: Single dose-group A
- 10 mg/kg or placebo iv (Other)
  Interventions: Biological: Single dose-group A
- 0.3 mg/kg or placebo sc (Other)
  Interventions: Biological: Single dose-group A; Biological: Multiple dose-Group B
- 0.1 mg/kg or placebo iv (multiple dose) (Other)
  Interventions: Biological: Multiple dose- Group B
- 0.3 mg/kg or placebo iv (multiple dose) (Other)
  Interventions: Biological: Multiple dose- Group B
- 3.0 mg/kg or placebo iv (Other)
  Interventions: Biological: Multiple dose- Group B
- 0.1 mg/kg or placebo sc (Other)
  Interventions: Biological: Multiple dose- Group B
- 0.3 mg/kg or placebo sc (multiple dose) (Other)
  Interventions: Biological: Multiple dose-Group B

INTERVENTIONS:
Biological: Single dose-group A — PF-00547659, single iv dose
  Arms: 0.03 mg/kg or placebo iv
Biological: Single dose-group A — PF-00547659, single iv dose
  Arms: 0.1 mg/kg or placebo iv
Biological: Multiple dose- Group B — PF-00547659, multiple dose
  Arms: 0.1 mg/kg or placebo iv (multiple dose)
Biological: Single dose-group A — PF-00547659, single iv dose
  Arms: 0.3 mg/kg or placebo iv
Biological: Multiple dose- Group B — PF-00547659, multiple dose
  Arms: 0.3 mg/kg or placebo iv (multiple dose)
Biological: Single dose-group A — PF-00547659, single dose
  Arms: 1.0 mg/kg or placebo iv
Biological: Single dose-group A — PF-00547659, single dose
  Arms: 3.0 mg/kg or placebo sc
Biological: Single dose-group A — PF-00547659, single dose
  Arms: 10 mg/kg or placebo iv
Biological: Single dose-group A — PF-00547659, single dose
  Arms: 0.3 mg/kg or placebo sc
Biological: Multiple dose-Group B — PF-00547659, multiple dose
  Arms: 0.3 mg/kg or placebo sc
Biological: Multiple dose- Group B — PF-00547659, multiple dose
  Arms: 0.1 mg/kg or placebo iv
Biological: Multiple dose- Group B — PF-00547659, multiple dose
  Arms: 0.3 mg/kg or placebo iv
Biological: Multiple dose- Group B — PF-00547659, multiple dose
  Arms: 3.0 mg/kg or placebo iv
Biological: Multiple dose- Group B — PF-00547659, multiple dose
  Arms: 0.1 mg/kg or placebo sc
Biological: Multiple dose-Group B — PF-00547659, multiple dose
  Arms: 0.3 mg/kg or placebo sc (multiple dose)

SUMMARY:
study to investigate the safety and efficacy properties of PF-00547659 in patients with active ulcerative colitis

ELIGIBILITY:
Inclusion Criteria:

* A positive histological diagnosis of UC ≥3 months prior to entry into the study. If a histological diagnosis is not available but all signs and symptoms suggest UC, the subject's eligibility should be discussed with Pfizer.
* Active UC as defined by a score of ≥6 on the Mayo score.
* An endoscopic (by flexible sigmoidoscopy) sub-score of ≥2 on the Mayo score determined within 7 days of first dosing.

Exclusion Criteria:

* Subjects with UC, which is confined to a proctitis on a flexible sigmoidoscopy.
* Subjects who have had surgery as a treatment for UC or are likely to require surgery within the duration of the study.
* Subjects displaying clinical signs of ischemic colitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety and toleration | up to 12 weeks
Endoscopic score changes as calculated using section 3 of the Mayo Score | up to 12 weeks
Disease activity score changes as calculated using the Mayo Score | up to 12 weeks

SECONDARY OUTCOMES:
Plasma concentrations of PF-00547659 | up to 12 weeks
Fecal concentrations of calprotectin | up to 12 weeks
Plasma concentrations of CRP | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Czechia (2):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- Pfizer Investigational Site, Aarhus C, Denmark
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Kiel
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Regensburg
- Pfizer Investigational Site, Oslo, Norway
- Pfizer Investigational Site, Nitra, Slovakia
- Spain (4):
  - Pfizer Investigational Site, Barcelona, BARCELONA
  - Pfizer Investigational Site, L'hospitalet DEL Llobregat, BARCELONA
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Majadahonda, Madrid

REFERENCES:
- [Derived] Vermeire S, Ghosh S, Panes J, Dahlerup JF, Luegering A, Sirotiakova J, Strauch U, Burgess G, Spanton J, Martin SW, Niezychowski W. The mucosal addressin cell adhesion molecule antibody PF-00547,659 in ulcerative colitis: a randomised study. Gut. 2011 Aug;60(8):1068-75. doi: 10.1136/gut.2010.226548. Epub 2011 Feb 11. PMID 21317177
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7281001&StudyName=A%20Study%20To%20Investigate%20The%20Safety%20And%20Efficacy%20Properties%20Of%20PF-00547659%20In%20Patients%20With%20Active%20Ulcerative%20Colitis